CLINICAL TRIAL: NCT03452358
Title: Clinical Evaluation of Partial Ceramic Posterior Restorations Cemented Using Immediate Dentin Sealing - a (#) Year Follow up From a Retrospective Study.
Brief Title: Survival Rate of Lithium Disilicate Crowns
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Carline van den Breemer, Principal Investigator, University Medical Center Groningen
Other Study IDs: 201500391
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Survival; Immediate Dentin Sealing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Partial Ceramic Indirect restoration — Placement of an partial ceramic indirect restoration with the use of immediate dentin sealing as an adjunct to adhesive cementation.
  Other Names: Immediate Dentin Sealing

SUMMARY:
A retrospective clinical study will be performed evaluating a large number of partial ceramic restorations (IPS e-Max press, Ivoclar, Liechtenstein) placed in general practice. Evaluation will be based on the well established Hickel criteria (Hickel et al, 2010). Rationale: IPS-e-max press has been made available to the market since 2006. Although millions of these restorations have been placed worldwide, clinical data are available of less than 200 single restorations only, covering observation periods of 2-8 years.(Guess et al, 2009; Etman en Woolford, 2010; Gehrt et al, 2012; Esquivel-Upshaw et al, 2012).

Objective: Study the survival of lithium disilicate restorations during regular check-ups in a private dental practice.

DETAILED DESCRIPTION:
Study the survival of lithium disilicate restorations during regular check-ups in a private dental practice. All included patients were followed-up with special emphasis on the partial restoration(s), every time they visited the dental practice for regular dental check-ups between 2015 and 2017. To assess these restorations a light photograph with a digital camera (Nikon (D7100, 60mm lens), Nikon, Amsterdam, The Netherlands) and an x-ray were taken from the partial posterior crowns and evaluated according to the modified United States Public Health Service (USPHS) criteria.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a patient must received one or more lithium disilicate restorations between 2006 and today.

Exclusion Criteria:

* No patients will be excluded from the study.

Age Groups: Child, Adult, Older Adult
Study Population: Patients participating in this study will be recruited from the patient population of the private dental practice 'Buijs tandartsen' in Groningen, the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Survival rate | from 2006 to 2018

SECONDARY OUTCOMES:
Quality of survival | from 2006 to 2018
  according to Hickel

IPD SHARING:
Plan to Share IPD: No